CLINICAL TRIAL: NCT05241353
Title: A Randomized Pilot Trial of a Tailored, Reduced-Frequency Approach to Dietary Self-Monitoring for Weight Loss
Brief Title: Project THRIVE: Evaluating Different Approaches to Dietary Self-Monitoring for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROJECTTHRIVE
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two arms (standard versus reduced-frequency). Participants will be assigned in a one-to-one fashion at baseline to one of the two groups.
Who Masked: Outcomes Assessor
Masking Description: Randomization will be concealed from outcome assessors. The allocation sequence will also be blinded in advance from individuals involved in the randomization process. However, it will not be fully possible to blind participants due to the nature of the trial (i.e., assignments will be evident to participants).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Self-Monitoring Group (Active Comparator): Standard behavioral treatment with a standard (full-frequency) self-monitoring prescription.
  Interventions: Behavioral: Full-Frequency Self-Monitoring; Behavioral: Standard Behavioral Treatment
- Reduced-Frequency Group (Experimental): Standard behavioral treatment with a reduced-frequency self-monitoring prescription.
  Interventions: Behavioral: Reduced Frequency Self-Monitoring; Behavioral: Standard Behavioral Treatment

INTERVENTIONS:
Behavioral: Reduced Frequency Self-Monitoring — Participants will be asked to record only a subset of daily eating throughout the intervention, with the prescription for self-monitoring individually tailored at baseline dependent on participants' self-reported eating patterns.
  Arms: Reduced-Frequency Group
Behavioral: Full-Frequency Self-Monitoring — Participants will be asked to record all contents of their diet throughout the intervention.
  Arms: Standard Self-Monitoring Group
Behavioral: Standard Behavioral Treatment — Participants will receive four individual coaching calls over 12 weeks. During coaching calls, participants will receive guidance on lowering calorie intake, increasing physical activity and use of specific behavioral strategies to increase the probability of success with weight loss.

SUMMARY:
This randomized pilot trial will compare two approaches to dietary self-monitoring for weight loss in the context of a low-intensity, remotely-delivered lifestyle modification program. Participants (N=40) will be randomized to perform detailed self-monitoring of all food and drink consumed each day or a reduced frequency, partial prescription involving recording only a subset of daily intake. The investigators will compare differences in weight loss as well as on relevant mechanistic, behavioral outcomes between groups at 12 weeks.

DETAILED DESCRIPTION:
Most lifestyle modification programs for weight loss require comprehensive, precise dietary self-monitoring (DSM) of all food and drink consumed each day. Although theoretically, such approaches should maximize the ability to identify dietary modifications leading to weight loss, the high level of burden associated with these requirements may produce suboptimal weight loss outcomes for many individuals by compromising DSM compliance, accuracy, and utilization for behavior change. A few prior trials have attempted to address this concern by relaxing the standard DSM requirement to record caloric intake precisely. However, such approaches are likely limited in efficacy because they reduce the utility DSM for implementing specific dietary changes. An alternative, as-of-yet untested approach to lower DSM burden would be to require that DSM be performed precisely but with reduced frequency, i.e., only during eating occasions strongly associated with eating patterns that threaten weight control. Thus, the purpose of the current pilot trial will be to compare the standard DSM protocol to a novel, reduced-frequency DSM approach in the context of a 12-week, low-intensity weight loss intervention. Participants (N = 40) will be randomized to receive either standard DSM advice or a reduced-frequency prescription and will receive four remotely-delivered individual coaching calls. The primary aim will be to investigate whether relative to standard DSM, reduced-frequency DSM can yield superior outcomes on four prospective indicators of long-term weight loss success (attitudes, DSM accuracy, utilization of DSM, and sustained compliance with DSM) and also produce comparable weight outcomes by 12 weeks.

All participants will receive a 12-week, low-intensity coaching-based intervention consisting of four individual coaching contacts. All study contacts will occur remotely using the HIPAA-compliant Zoom service at Drexel University. Participants will first complete preliminary eligibility screening via telephone and eligibility will be confirmed during an individual baseline assessment, during which participants will also receive an overview of study procedures. Following the baseline assessment but prior to the first coaching call, participants will engage in fully comprehensive, standard DSM for one week to generate data on the participant's typical dietary patterns, and these data will be used to tailor the DSM prescription in the reduced-frequency DSM group. Participants will also be provided with weekly electronic reading material on principles of behavioral weight control. The first coaching call will be one hour in duration and will provide an overview of general behavioral principles of weight control, including requiring the participant to set specific calorie reduction, self-monitoring and physical activity goals. Participants will also be randomized at during the first coaching call one-to-one fashion to either receive standard DSM advice or to receive a reduced frequency prescription that requires recording only a subset of eating each day throughout the intervention. Permuted block randomization will be performed, stratified on baseline BMI (groups: BMI <30, BMI 30-35, BMI >35). Depending on the participant's assignment, he/she/they will be assigned during the baseline coaching call to either continue recording all dietary intake each day (using the Fitbit mobile application) or record a subset of eating tailored to the individual's within-day dietary patterns using a simple algorithm. Subsequent coaching calls will focus on a review of adherence to dietary and physical activity goals and problem-solving solutions to the participant's stated barriers to adherence. Participants in the reduced-frequency group will also have opportunities to modify the self-monitoring prescription during subsequent coaching calls depending on the perceived feasibility of their current prescription. Lastly, participants in both groups will complete a post-treatment assessment during which self-report measures will be completed and skills to maintain after treatment will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Currently living in the United States
* Current body mass index (BMI) of 25-50 kg/m2, with individuals with BMI > 50 excluded due to the higher risk of medical complications
* Access to a regular internet connection
* Ability to understand and provide informed consent
* Individuals must provide consent for the research team to contact their personal physician if necessary, to provide clearance or to consult about rapid weight loss
* Proficiency in speaking, reading, and writing English
* Ability to engage in physical activity, defined as the ability to walk at least the length of two city blocks without stopping
* Access to or willing to purchase a digital wireless body weight scale

Exclusion Criteria:

* Present involvement in another lifestyle modification or obesity treatment program
* Currently breastfeeding, pregnant or planning to become pregnant within 4 months from the time of screening
* Having lost more than 5% of body weight in the past 3 months
* History of bariatric surgery
* Acute suicide risk (exclude if present in the past 2 weeks or if any attempts were made in past 2 years)
* Self-reported diagnosis of a medical or psychiatric condition that could make standard behavioral weight loss treatment contraindicated, including: insulin-dependent diabetes (type 1 or type 2; individuals with diabetes who do not take insulin will not be excluded), cancer, loss-of-control eating (three or more times in the past month), inappropriate compensatory behaviors to control weight (vomiting, misuse of laxatives or diuretics, or compelled exercise) in the past month, current unmedicated bipolar or psychotic disorder, or current psychiatric symptoms that would interfere with an individual's ability to complete the program.
* Technological or interpersonal difficulties contraindicating participation in a remotely delivered coaching program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Percent Weight Loss at Week 12 | Week 0 (Baseline), Week 12 (Post-Treatment)
  Weight will be assessed at baseline and weekly throughout the intervention. Participants will be instructed to self-weigh on one consistent morning per week before 11am, following specific instructions (i.e., wear light clothing, keep scale on a flat surface, weigh before eating or drinking) and then self-report weight using the Fitbit app where it can be later exported by research staff. Participants will be required to self-weigh using a reliable, digital wireless scale that can estimate weight to the nearest tenth of a pound. Percent weight loss at week 12 will be calculated as the percentage loss in initial body weight at baseline by the time of the post-treatment assessment.

SECONDARY OUTCOMES:
Perceived Autonomy Support at Week 12 | Week 12 (Post-Treatment)
  Perceived autonomy support will be evaluated using a modified version of the Health Care Climate Questionnaire, which has strong psychometric properties (α = 0.97). This 15-item measure examines the extent to which an individual feels supported by their health care provider to take personal responsibility for his or her health. Scores are calculated as the mean of all items on the scale, reverse-scoring item 13. Scores on the scale range from 1 to 7, with higher scores indicating higher perceived autonomy support. Perceived autonomy support will be assessed only at post-treatment.
Change in Weekly Compliance with DSM from Weeks 1 to 12 | Week 1 through Week 12 (Post-Treatment)
  Compliance with dietary self-monitoring (DSM) will be operationalized as the proportion of required meals and snacks recorded (based on the participant's eating plan) each week. Recording of a given meal or snack will be defined as the presence of at least one food item logged for a snack and two food items logged for a meal. To calculate the proportion of required meals and snacks recorded each day, the total number of recorded meals and snacks will be divided by a constant representing the "expected" number of eating occasions (two for the reduced frequency DSM group; for the standard DSM group, this value will correspond to the number of eating occasions in the participant's eating plan). This proportion will initially be computed at the day level and will then be averaged across each week during the intervention phase for each participant. Change in compliance with DSM will be evaluated weekly over the course of the 12-week intervention (i.e., weeks 1-12).
Change in Week 3 Utilization of Strategies to Ensure DSM Accuracy at Week 12 | Week 3, Week 12 (Post-Treatment)
  This variable will be assessed via self-report at week 3 and at post-treatment (Week 12). Participants will be asked to rate on a five-item Likert scale the extent to which 10 statements describing efforts to perform highly precise DSM (e.g., "I always tracked hidden calories like oils, cream, butter, and added sugars," "I always weighed or measured my food before entering it into my food record") have applied to them over the past three weeks (1 = Never, 5 = Always). A composite score will be computed as the mean score of all items on the scale. Change in this variable will be assessed as a difference score between week 3 and post-treatment.
Change in Week 3 Utilization of DSM for Dietary Change at Week 12 | Week 3, Week 12 (Post-Treatment)
  Utilization of DSM will first be assessed at week 3, to ensure that participants have first had an opportunity to fully engage in DSM for several weeks, and then again at post-treatment. This measure will ask participants to rate the extent to which they utilized self-monitoring records to make specific dietary changes over the past three weeks. Participants will be presented with a list of 15 potential dietary modifications related to weight control (e.g., decreased intake of calories from beverages, increased consumption of fruits/vegetables) and asked to endorse which, if any, they have made related to their personal DSM practice during the intervention. A total score for utilization of DSM will be computed as the total number of items on the list endorsed. Change in this variable will be assessed as a difference score between week 3 and post-treatment (week 12).
Change in Baseline Attitudes Towards DSM at Week 12 | Week 0 (Baseline), Week 12 (Post-Treatment)
  Attitudes towards DSM will be assessed at baseline (Week 0) and post-treatment (Week 12) using four, five-point custom Likert scale items. Items will assess participant perceptions of usefulness ("I think that tracking my calories is useful for losing weight"), liking ("I like tracking what I eat using the Fitbit app"), burden associated with DSM ("Tracking my calories feels like too much work to be worth it") and intention to continue engaging in DSM over the upcoming year (1 = not at all confident, 5 = extremely confident). A composite index of attitudes towards DSM will be computed from the average of the perceived usefulness, liking, burden, and intention to maintain items, reverse-scoring the burden item. Change in attitudes towards DSM will be assessed as a difference score between baseline and post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University Center for Weight, Eating & Lifestyle Science, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No